CLINICAL TRIAL: NCT05929040
Title: Using the Behaviour Change Technique Taxonomy v1 to Conceptualize the Clinical Content of a Preliminary Randomised Controlled Study of an Online Mindfulness-based Cognitive Intervention for Chemsex
Brief Title: The Use of Cognitive Mindfulness for Chemsex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Metropolitan University (Other)
Responsible Party: Principal Investigator, Samantha Banbury, Dr Samantha Banbury, London Metropolitan University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: London Met University
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Substance Use
Keywords: Chemsex; Cognitive mindfulness; Sexual self efficacy; Well-being
MeSH Terms: conditions — Substance-Related Disorders; Chemsex

STUDY DESIGN:
Intervention Model Description: Waitlist control. An experimental group and a delayed group over 8 weeks Waitlist controlled RCT (N= 16 immediate group, N=15)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate group (Experimental): Randomized controlled waitlist study
  Behavioral: Mindfulness based cognitive intervention based on the behavioural change techniques taxonomy
  An online mindful cognitive intervention is used as a proposed treatment intervention for chemsex among men ho have sex with men in the United Kingdom.
  Interventions: Behavioral: mindful cognitive intervention
- Delayed group (Other): Randomized controlled waitlist study
  Behavioral: Mindfulness based cognitive intervention based on the behavioural change techniques taxonomy
  An online mindful cognitive intervention is used as a proposed treatment intervention for chemsex among men who have sex with men in the United Kingdom.
  Interventions: Behavioral: mindful cognitive intervention

INTERVENTIONS:
Behavioral: mindful cognitive intervention — Mindfulness based cognitive intervention based on the behavioural change techniques taxonomy

SUMMARY:
Title of research: A preliminary RCT of an online mindfulness-based cognitive intervention for Chemsex

Research aim: To determine how an online mindfulness-based cognitive intervention, might reduce Chemsex engagement, risky sexual behaviours, sexual self-efficacy and increase overall wellbeing among men who have sex with men.

Research intention: If the mindfulness based cognitive intervention reduces Chemsex engagement and risky sexual behaviours and supports sexual and general wellbeing, then we would repeat this study on a larger scale within the National Health Service among men who have sex with other men and who engage in Chemsex. Both academic output and dissemination accordingly.

A brief overview of intervention:

Chemsex, sometimes coined as Chemfun, is a term used to describe the use of psychoactive substances with the intention of enhancing and/or facilitating the sexual experience/arousal and predominates among gay and bisexual men. Chemsex drugs tend to include, γ-hydroxybutyric acid and congeners, methamphetamine, mephedrone, erectile dysfunction agents, and alkyl nitrites often in combination.

A growing body of research has suggested that mindfulness supports minimize drug using behaviors HIV stress and risky sexual behaviours. However, there appears no current mindfulness intervention that has been evidenced for Chemsex. Our intervention is hoped to become part of a multidisciplinary approach in supporting Chemsex which includes a cross-over effect between drugs, sexual well-being, and general wellbeing.

Quantitatively, the research is structured so that participants will be randomized to either the experimental or control group (n=20 experimental; n=20 control waitlist). The MBCI for each group is 1 month (4 wks experimental and 4 wks waitlist control). This is followed by a 3-month follow-up to determine the sustainability of this intervention. Qualitatively, participants will be asked approx 8 open-ended feedback questions forming part of 4 groups of 10, at the 3-month follow-up.

DETAILED DESCRIPTION:
The principal researcher developed an online cognitive mindfulness intervention.

The main target in this study was to engage participants with mindfulness exercises whilst improving wellbeing and mindfulness whilst reducing Chemsex use. The main exercises included mindfulness, breathing exercises, relaxation techniques, being mindful of the senses and the body and understanding of the self. This online mindfulness based cognitive intervention contains cognitive, emotional, and behavioural factors and each of the 4 sessions included substance use and sexual behaviour, working with the inner critic and high-risk situations, sex without drugs and sexual identity and psychosexual wellbeing, substance use and self-compassion. Homework exercises were encouraged which consisted of education, training, modelling, and enablement. To expand, education included psychoeducational information on chemsex, sexual wellbeing, and mindfulness along with additional resources. Training provided the instructions on how to go about engaging in these online activities. Modelling provides examples in action such as MSM discussing their experiences of Chemsex including verbal persuasion and challenging negative self-talk, and how to go about doing the exercises, and enablement is aimed at increasing participants capability of engaging in these activities towards wellbeing. This would be further supported by charts, self-monitors, diaries, and journaling. Further, prompts, action plans, and cues were supportive intervention components. Feedback and support along with discussing the educational components, training, modelling and enablement had been addressed throughout the duration of this study.

The development of the mindfulness based cognitive intervention has been based on a behavioral change techniques taxonomy. This have been used because the behavioural change techiques taxonomy has been rigorously tested to evidence the effectiveness in support of interventions associated with change behaviour. The 93 behavior change techniques are the active ingredients of behavior change where each intervention is likely to consist of more than one behaviour change technique and serve as having more than one function. In total, the intervention in this study included 15 domains in which 35 out of the 93 behaviour change techniques listed in the behavioural change technique taxonomy were identified. The selection of these domains used a process of triangulation to ensure consistency in mapping the behaviour change techniques to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old and above
* Are engaged in chemsex
* Men who have sex with men
* Can read and write English
* Had access to a password-protected laptop/computer
* Registered with a General Practitioner
* Registered with a health care service supporting substance use/chemsex.

Exclusion Criteria:

* Aged below 18 years old
* Those who do not engage in Chemsex
* Are not registered with a General Practitioner
* Did not have access to a password-protected laptop/computer
* Are not registered with a health care service supporting substance use/chemsex
* Have difficulties reading and writing in English

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — men who have sex with men
Enrollment: 29 (Actual)
Dates: Start 2022-03-05 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Changes in Chemsex behaviour, measurements taken at weeks 0, 8 and 12 | Measurements taken at weeks 0, 8 and 12
  There is currenlty no standardised questionnaire on chemsex. This is a 19-item questionnaire with 4 response categories (1=never through to 4= always). Scores ranged between 19 (low chemsex engagement) to 76 (very high chemsex engagement). 19 No Chemsex; 20-34 Low chemsex; 35-50 Moderate chemsex; 51- 66 High chemsex and 67 + very high chemsex. Questions 1-4 includes drug use, 5-7 self-care, 8-10 lifestyle, 11-14 risk behaviour, 15-19 well-being/mental health.
Changes in cognitive mindfulness, measurements taken at weeks 0, 8 and 12. | Measurements taken at weeks 0,8 and 12
  The Cognitive and Affective Mindfulness Scale-Revised. This is a 10-item measure with four response categories 1= rarely/not at all to 4 = almost always. Higher scores indicate higher levels of mindfulness (range 4-40). Cronbach's alphas ranged between 0.82 and 0.84.
Changes in sexual self efficacy, measurements taken at weeks 0, 8 and 12. | Measurements taken at weeks 0, 8 and 12
  This is a six-item questionnaire which consists of 4 response categories (1=not at all through to 4= very much). Cronbach's alpha ranges between 0.58- 0.74. Questions centre on the self-efficacy for carrying out healthy sexual behaviours including condom use and sexual consent. There is no reverse scoring. Scores range from 6 (little to no self-efficacy) to 24 (high self-efficacy). This will be adapted accordingly… Think about the time you have engaged in chemsex, how confident are you that you could..
Changes in wellbeing, measurements taken at weeks 0, 8 and 12. | Measurements taken at weeks 0, 8 and 12
  This is a positively worded 7 item questionnaires with 5 response categories looking at functioning and feeling aspects of well-being. The response categories include 1=none of the time to 5=all of the time. Cronbach alpha- 0.89-0.91. There is no reverse scoring. Scores range from 7 to 35 where the latter is the highest level of wellbeing.

CONTACTS AND LOCATIONS:
Locations (1):
- Samantha Banbury, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alvy LM, McKirnan DJ, Mansergh G, Koblin B, Colfax GN, Flores SA, Hudson S; Project MIX Study Group. Depression is associated with sexual risk among men who have sex with men, but is mediated by cognitive escape and self-efficacy. AIDS Behav. 2011 Aug;15(6):1171-9. doi: 10.1007/s10461-010-9678-z. PMID 20217471
- [Result] Flores Anato JL, Panagiotoglou D, Greenwald ZR, Trottier C, Vaziri M, Thomas R, Maheu-Giroux M. Chemsex practices and pre-exposure prophylaxis (PrEP) trajectories among individuals consulting for PrEP at a large sexual health clinic in Montreal, Canada (2013-2020). Drug Alcohol Depend. 2021 Sep 1;226:108875. doi: 10.1016/j.drugalcdep.2021.108875. Epub 2021 Jun 25. PMID 34218004
- [Result] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Result] Banbury, S., Moneta, G & Chandler, C (2021) An exploratory study examining the relationship between sexual self efficacy and premature ejaculation mediated by depression, anxiety and sexual fantasy among a British cohort. Sexual and Relationship Therapy, (7), 1-17DOI: 10.1080/14681994.2021.1932796
- [Result] Banbury, S., Lusher, J., Snuggs, S & Chandler, C., (2021). Mindfulness-based therapies for men and women with sexual dysfunction: a systematic review and meta-analysis. Sexual and Relationship Therapy, DOI: 10.1080/14681994.2021.1883578.
- [Result] Bohn A, Sander D, Kohler T, Hees N, Oswald F, Scherbaum N, Deimel D, Schecke H. Chemsex and Mental Health of Men Who Have Sex With Men in Germany. Front Psychiatry. 2020 Nov 4;11:542301. doi: 10.3389/fpsyt.2020.542301. eCollection 2020. PMID 33329083
- [Result] Bandura, A. (1992). Exercise of personal agency through the self-efficacy mechanism. In R. Schwarzer (Ed.), Self-efficacy (pp.3-38). Washington DC US: Hemisphere Publishing Corp.
- [Result] Bandura, A., (1997). Self-efficacy: The exercise of control. New York: W. H. Freeman. ISBN 978-0- 7167- 2850-4. ISBN 0-7167-2850-8, OCLC 36074515
- [Result] Blomquist PB, Mohammed H, Mikhail A, Weatherburn P, Reid D, Wayal S, Hughes G, Mercer CH. Characteristics and sexual health service use of MSM engaging in chemsex: results from a large online survey in England. Sex Transm Infect. 2020 Dec;96(8):590-595. doi: 10.1136/sextrans-2019-054345. Epub 2020 Mar 5. PMID 32139497
- [Result] Bossio JA, Basson R, Driscoll M, Correia S, Brotto LA. Mindfulness-Based Group Therapy for Men With Situational Erectile Dysfunction: A Mixed-Methods Feasibility Analysis and Pilot Study. J Sex Med. 2018 Oct;15(10):1478-1490. doi: 10.1016/j.jsxm.2018.08.013. PMID 30297094
- [Result] Bowen S, Enkema MC. Relationship between dispositional mindfulness and substance use: findings from a clinical sample. Addict Behav. 2014 Mar;39(3):532-7. doi: 10.1016/j.addbeh.2013.10.026. Epub 2013 Oct 29. PMID 24290208
- [Result] Bracchi M, Stuart D, Castles R, Khoo S, Back D, Boffito M. Increasing use of 'party drugs' in people living with HIV on antiretrovirals: a concern for patient safety. AIDS. 2015 Aug 24;29(13):1585-92. doi: 10.1097/QAD.0000000000000786. PMID 26372268
- [Result] Cadogan CA, Ryan C, Francis JJ, Gormley GJ, Passmore P, Kerse N, Hughes CM. Development of an intervention to improve appropriate polypharmacy in older people in primary care using a theory-based method. BMC Health Serv Res. 2016 Nov 16;16(1):661. doi: 10.1186/s12913-016-1907-3. PMID 27852287
- [Result] Cane J, O'Connor D, Michie S. Validation of the theoretical domains framework for use in behaviour change and implementation research. Implement Sci. 2012 Apr 24;7:37. doi: 10.1186/1748-5908-7-37. PMID 22530986
- [Result] Carrico AW, Neilands TB, Dilworth SE, Evans JL, Gomicronmez W, Jain JP, Gandhi M, Shoptaw S, Horvath KJ, Coffin L, Discepola MV, Andrews R, Woods WJ, Feaster DJ, Moskowitz JT. Randomized controlled trial of a positive affect intervention to reduce HIV viral load among sexual minority men who use methamphetamine. J Int AIDS Soc. 2019 Dec;22(12):e25436. doi: 10.1002/jia2.25436. PMID 31860172
- [Result] Chan, K.K.S., Lee, C.W.L., & Mak, W.W.S., (2018). Mindfulness model of stigma resistance among individuals with psychiatric disorders. Mindfulness, 9(5), 1433-1442. http://dx.doi.org/10.1007/s12671- 018-0887-2
- [Result] Dakwar E, Nunes EV, Hart CL, Foltin RW, Mathew SJ, Carpenter KM, Choi CJJ, Basaraba CN, Pavlicova M, Levin FR. A Single Ketamine Infusion Combined With Mindfulness-Based Behavioral Modification to Treat Cocaine Dependence: A Randomized Clinical Trial. Am J Psychiatry. 2019 Nov 1;176(11):923-930. doi: 10.1176/appi.ajp.2019.18101123. Epub 2019 Jun 24. PMID 31230464
- [Result] Giorgetti R, Tagliabracci A, Schifano F, Zaami S, Marinelli E, Busardo FP. When "Chems" Meet Sex: A Rising Phenomenon Called "ChemSex". Curr Neuropharmacol. 2017;15(5):762-770. doi: 10.2174/1570159X15666161117151148. PMID 27855594
- [Result] Gu J, Strauss C, Bond R, Cavanagh K. How do mindfulness-based cognitive therapy and mindfulness-based stress reduction improve mental health and wellbeing? A systematic review and meta-analysis of mediation studies. Clin Psychol Rev. 2015 Apr;37:1-12. doi: 10.1016/j.cpr.2015.01.006. Epub 2015 Jan 31. PMID 25689576
- [Result] Kurtz SP. Post-circuit blues: motivations and consequences of crystal meth use among gay men in Miami. AIDS Behav. 2005 Mar;9(1):63-72. doi: 10.1007/s10461-005-1682-3. PMID 15812614
- [Result] Maxwell S, Shahmanesh M, Gafos M. Chemsex behaviours among men who have sex with men: A systematic review of the literature. Int J Drug Policy. 2019 Jan;63:74-89. doi: 10.1016/j.drugpo.2018.11.014. Epub 2018 Dec 1. PMID 30513473
- [Result] McKirnan DJ, Ostrow DG, Hope B. Sex, drugs and escape: a psychological model of HIV-risk sexual behaviours. AIDS Care. 1996 Dec;8(6):655-69. doi: 10.1080/09540129650125371. PMID 8993716
- [Result] Rostosky SS, Dekhtyar O, Cupp PK, Anderman EM. Sexual self-concept and sexual self-efficacy in adolescents: a possible clue to promoting sexual health? J Sex Res. 2008 Jul-Sep;45(3):277-86. doi: 10.1080/00224490802204480. PMID 18686156
- [Result] Tomkins A, George R, Kliner M. Sexualised drug taking among men who have sex with men: a systematic review. Perspect Public Health. 2019 Jan;139(1):23-33. doi: 10.1177/1757913918778872. Epub 2018 May 30. PMID 29846139